Measuring the effect of using the Arabic Otago Exercise Program on falls and falls-related factors

in People with Multiple Sclerosis

Date: March 23rd, 2021

NCT number: not assigned yet.

Statistical analysis

Demographics and health-related information will be presented using mean and

standard deviation as well as frequency statistics. ANOVA statistics will be used to calculate

the mean differences between and within groups. Statistical Package for the Social Sciences

(SPSS) 23.0 (SPSS®: Inc., Chicago, IL, USA) will be used to analyze the results of the study.

A priori power analysis was conducted using the software package, GPower (Faul,

Erdfelder, Buchner, & Lang, 2009) with a power of 0.8 and an alpha of 0.05 and an effect size

of 0.8 for balance (Gunn, Markevics, Haas, Marsden, & Freeman, 2015). The analysis

indicated that a total sample size of 42 participants in both groups (21 in each group) would be

sufficient to evaluate the mean difference between groups. However, 50 participants will be

recruited to take into considerations drop out incidences.